CLINICAL TRIAL: NCT03691493
Title: A Phase II Multi-Institutional Study of Concurrent Radiotherapy, Palbociclib, and Hormone Therapy for Treatment of Bone Metastasis in Breast Cancer Patients
Brief Title: Radiation Therapy, Palbociclib, and Hormone Therapy in Treating Breast Cancer Patients With Bone Metastasis
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Mylin Torres, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00105944; NCI-2018-02000 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4472-18 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Estrogen Receptor Positive; HER2/Neu Negative; Metastatic Breast Carcinoma; Metastatic Malignant Neoplasm in the Bone; Progesterone Receptor Positive; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Fulvestrant; Letrozole; palbociclib; Radiotherapy; Radiation; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Radiation, palbociclib, hormone therapy (Experimental): Patients undergo radiation therapy over 5-10 days and receive palbociclib PO QD on days 1-21. At the discretion of treating physician, patients also receive letrozole, anastrozole, exemestane, or tamoxifen PO QD on days 1-28, or fulvestrant IM on days 1 and 15 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant; Drug: Letrozole; Drug: Palbociclib; Radiation: Radiation Therapy; Drug: Tamoxifen

INTERVENTIONS:
Drug: Anastrozole — Given PO
  Other Names: Arimidex; ICI D1033; ZD-1033
Drug: Exemestane — Given PO
  Other Names: Aromasin; FCE-24304
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; ICI 182,780; ZD9238
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Palbociclib — Given PO
  Other Names: Ibrance; PD-0332991
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiation; Radiation; Radiotherapeutics
Drug: Tamoxifen — Given PO
  Other Names: Soltamox; Nolvadex

SUMMARY:
This phase II trial studies how well radiation therapy given with standard care palbociclib and hormone therapy work in treating patients with breast cancer that has spread from one part of the body to the bone. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Palbociclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Antihormone therapy, such as fulvestrant, letrozole, anastrozole, exemestane, or tamoxifen, may lessen the amount of estrogen made by the body. Giving radiation therapy, palbociclib, and hormone therapy may work better in treating breast cancer patients with bone metastasis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the response rate three months post-conventionally fractionated radiotherapy, relative to baseline, for bone metastases in breast cancer patients receiving concurrent palbociclib and hormone therapy treatment.

SECONDARY OBJECTIVES:

I. To determine whether conventionally fractionated radiotherapy in combination with palbociclib and hormone therapy in breast cancer patients with bone metastases adversely increases the frequency and severity of palbociclib toxicities including grade 3 neutropenia.

II. To determine whether radiotherapy in combination with palbociclib in breast cancer patients with bone metastases adversely increases the frequency and severity of radiotherapy toxicities including neurological and bone injury.

III. To assess fatigue, quality of life, and depression before and after radiotherapy for bone metastases in metastatic breast cancer patients treated with palbociclib.

IV. To determine progression free survival (PFS) and overall survival (OS) in breast cancer patients treated with palbociclib and concurrent radiotherapy to bone metastases.

V. To evaluate the relationship between volume of irradiated bone and side effects of treatment, including leukopenia and neutropenia.

TRANSLATIONAL RESEARCH OBJECTIVES:

I. To collect, store, and analyze circulating tumor-derived deoxyribonucleic acid (ctDNA) in metastatic breast cancer patients treated with palbociclib and radiotherapy to bone metastases and to determine the relationship between ctDNA and responders versus non-responders, PFS, and OS.

II. To collect, store, and analyze plasma for inflammatory cytokine measurements and determine their relationship with fatigue, depression, and quality of life before and after radiotherapy for bone metastases in metastatic breast cancer patients treated with palbociclib.

III. To collect, store, and analyze ribonucleic acid (RNA) for gene expression to identify functional biology processes over-represented in genes differentially regulated among patients who develop toxicities versus those who do not and those who are responders versus those who are not and to identify transcriptional regulatory pathways driving observed differences in gene expression.

OUTLINE:

Patients undergo conventional radiation therapy over 5-10 days and receive palbociclib orally (PO) once daily (QD) on days 1-21. At the discretion of treating physician, patients also receive letrozole, anastrozole, exemestane, or tamoxifen PO QD on days 1-28, or fulvestrant intramuscularly (IM) on days 1 and 15 of cycles 1 and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 and 3 months.

ELIGIBILITY:
Patient Selection Guidelines:

* Patients must have the psychological ability and general health that permits completion of the study requirements and required follow up
* Women of childbearing potential who are sexually active should be willing and able to use medically acceptable forms of contraception during protocol treatment

Inclusion Criteria:

* Pathologically confirmed metastatic breast cancer
* Known estrogen, progesterone, and human epidermal growth factor receptor 2 (Her2) status of either primary tumor or metastasis
* Metastatic estrogen receptor positive (ER+) or progesterone receptor positive (PR+), Her2/neu negative breast cancer patients with imaging confirming bone metastasis within 60 days of radiation simulation
* Must be actively receiving palbociclib (125 or 100 mg PO daily for 3 weeks followed by a week off during 28-day cycles) plus one of the following hormone therapies for at least 28 days:

  * Fulvestrant (500 mg IM injection on days 1 and 15 cycle one and then on day one of each subsequent cycle (28 days) -or-
  * Letrozole (2.5 mg PO daily) -or-
  * Anastrozole (1 mg PO daily) -or-
  * Exemestane (25 mg PO daily) -or-
  * Tamoxifen (20 mg PO daily)
* Patients must be willing and able to provide written informed consent/assent for the trial
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Karnofsky performance status (KPS) ≥ 60% within 60 days prior to registration
* Must have bone disease that is either symptomatic (i.e. pain) or has a lytic or mixed lytic disease that can be assessed by computed tomography (CT), magnetic resonance imaging (MRI), bone scan or positron emission tomography (PET)/CT within 60 days prior to radiotherapy on this study
* One previous line of chemotherapy in advanced disease is allowed
* Appropriate stage for study entry based on the following diagnostic workup:

  * History and physical examination within 60 days prior to registration
  * Clinical grade CT scans of the chest, abdomen, and pelvis with radionuclide bone scan OR whole body PET/CT documenting metastatic disease prior to radiotherapy on this protocol or MRI documenting site of metastatic disease to be treated on protocol
* Patient must be eligible for palliative radiotherapy (conventional radiation either 30 Gy in 10 fractions or 20 Gy in 5 fractions) for up to 4 separate anatomic regions containing bone metastases defined by 4 separate and not overlapping radiation plans
* Absolute neutrophil count ≥ 1000/mcl (obtained within 14 days prior to registration on study)
* Platelets ≥ 75,000 mm³ (obtained within 14 days prior to registration on study)
* Hemoglobin ≥ 8.0 g/dl (obtained within 14 days prior to registration on study) (Note: The use of transfusion or other intervention to achieve hemoglobin [Hgb] ≥ 8.0g/dl is acceptable) (obtained within 60 days prior to registration on study)
* For females of child-bearing potential, negative serum or urine pregnancy test within 14 days prior to radiation simulation
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Prior Treatment:

  * Patients may or may not have received radiotherapy or neoadjuvant or adjuvant chemotherapy in the treatment of their initial, non-metastatic breast cancer, but must be entered on study after their last dose of radiotherapy, last cycle of chemotherapy and biologic therapy (if applicable) and have sufficient resolution of side effects per physician assessment at time of radiotherapy
  * Patients must have not active wound healing issues from surgery and sufficient resolution of surgical side effects, per physician assessment, at time of radiotherapy
  * If patients have one line of chemotherapy for advanced disease, patients must be entered on study after their last dose of chemotherapy and have sufficient resolution of side effects per physician assessment at time of radiotherapy
  * Patients must have already initiated palbociclib (3 weeks on, 1 week off) and hormone therapy for at least 28 days prior to radiotherapy
  * During radiotherapy, no other investigation or commercial agents or therapy for cancer other than palbociclib, bisphosphonates, rank ligand inhibitors, and hormone therapy should be administered
  * Patients may have received bisphosphonates or rank ligand inhibitors prior to enrollment on study

Exclusion Criteria:

* Co-existing or prior invasive non-breast malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years
* Previous radiation dose, date, fraction size, must be reported for prior invasive malignancy
* Previous palliative radiation to the disease to be treated on protocol (including radiopharmaceuticals)
* Patients prescribed stereotactic body radiation therapy (SBRT) for bone metastasis to be treated on this protocol will be excluded
* Metastases to be treated on protocol located within 2 cm from a previously irradiated structure:

  * Spinal cord previously irradiated to > 40 Gy (delivered in ≤ 3 Gy/fraction)
  * Brachial plexus previously irradiated to > 50 Gy (delivered in ≤ 3 Gy/fraction)
  * Small intestine, large intestine, or stomach previously irradiated to > 45 Gy (delivered in ≤ 3 Gy/fraction)
  * Brainstem previously irradiated to > 50 Gy (delivered in ≤ 3 Gy/fraction)
  * Whole lung previously irradiated with prior V20 Gy > 35% (delivered in ≤ 3 Gy/fraction)
* Untreated brain metastases or unstable/progressive brain metastases (imaging of treated brain metastases must be performed within 28 days of registration for this protocol to confirm brain metastases stability)
* Severe, active co-morbidity such as congestive heart failure (CHF) or unstable angina within last 6 months, transmural myocardial infarction within the last 6 months. Acute bacterial or fungal infection requiring intravenous (IV) antibiotics at time of registration, chronic obstructive pulmonary disease (COPD) or other respiratory illness requiring hospitalization at time of registration
* Lactating females must cease expression of milk prior to registration
* Temperature above 100.4° Fahrenheit
* Human immunodeficiency virus (HIV) positive with cluster of differentiation 4 (CD4) count < 200 cells/ microliter. HIV positive patients are eligible, provided they are receiving treatment with highly active antiretroviral therapy (HAART) and have a CD4 count > 200 cells/microliter within 28 days prior to registration. HIV testing is not required for eligibility for this protocol. This exclusion criteria is necessary because the treatments involved in this protocol may be significantly immunosuppressive
* Previous chemotherapy or radiotherapy within 2 weeks prior to registration or patients who have not recovered from adverse events due to previous chemotherapy and radiotherapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy. Indolent cancers (such as low risk prostate or In-Situ cancers) that are not being treated are acceptable
* Has active autoimmune disease that has required continued systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Cannot receive concurrent cytotoxic chemotherapy (e.g. taxanes, cytoxan, anthracyclines, platinum based aged, capecitabine) at time of registration or during radiation treatment on this study
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 90 days after the last dose of trial treatment
* Absolute neutrophil count < 1000/microliter (mcl)
* Platelets < 75,000 mm
* Hemoglobin < 8.0 g/dl
* Concurrent therapy with other investigational products is not allowed
* Receiving medications or substances that are potent inhibitors or inducers of cytochrome P450, family 3, subfamily A (CYP3A) isoenzymes, as palbociclib is primarily metabolized by CYP3A4 enzymes, within 7 days of registration:

  * Inhibitors - boceprevir, clarithromycin, indinavir, delavirdine, conivaptan, itraconazole, ketoconazole, lopinavir, mibefradil, miconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, suboxone, telaprevir, telithromycin, voriconazole, amprenavir, atazanavir, diltiazem, erythromycin, fosamprenavir, verapamil, and grapefruit, grapefruit juice or any product containing grapefruit
  * Inducers - carbamazepine, phenytoin, primidone, rifampin, rifapentine, St. John's wort, felbamate, nevirapine, phenobarbital, rifabutin
* Receiving hormone replacement therapy (e.g. topical estrogens, but not intra-vaginal preparations, raloxifene, megestrol acetate)
* Patients with clinical signs of cord compression, patients with radiographic evidence of cord compression are eligible for enrollment but cannot have clinical signs of cord compression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2022-10-13 (Actual); Study Completion 2022-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mylin Torres, MD, Principal Investigator — Emory University
Locations (10):
- United States (10):
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Maine Medical Center-Bramhall Campus, Portland, Maine

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Started | 36
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 24
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Count of participants
  Participants
    United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response rate will be estimated as the number of responders divided by the number of patients evaluated for response. Among patients who present with pain, responders will be considered those patients who have a 2 point decrease in the Brief Pain Inventory (BPI), and among those who do not present with pain (radiotherapy due to risk of unstable fracture or cord compression), responders will be considered those without development of a pathologic fracture or neurologic compromise (cord compression) due to cancer on imaging.
Time Frame: Up to 3 months post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 35
Participants
  Responders | 29
  Non-responders | 6

2. Secondary Outcome: Response Rate Incorporating BPI and Analgesic Measures According to International Bone Consensus Guideline Criteria
Description: Response rate will be estimated as the number of responders divided by the number of patients evaluated for response. Among patients who present with pain, responders will be considered those patients who fulfill the International Bone Consensus response criteria using the BPI item rating maximum pain over the last 3 days at the index site and analgesic usage for the treated site within the last 24 hours prior to assessment. Among patients who do not present with pain (radiotherapy due to risk of unstable fracture or cord compression), responders will be considered those without development of a new pathologic fracture or worsening neurologic compromise (cord compression) due to cancer on imaging.
Time Frame: Up to 3 months post radiation
Population: 27 participants were evaluable
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 27
Participants
  Responders | 18
  Non-responders | 2
  Intermediate | 7

3. Secondary Outcome: Number of Participants With Adverse Events Graded According to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: Adverse events, such as bone fracture following radiotherapy, any grade 3 toxicity (except neutropenia or leukopenia), grade 4 neutropenia, grade 4 leukopenia, grade 3 febrile neutropenia, or grade 3 brachial plexopathy or spinal cord injury, will be summarized descriptively.
Time Frame: Up to 3 months post radiation
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Participants | 31

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS will be estimated using the Kaplan-Meier method.
Time Frame: Up to 44 months post radiation
Measure: Median (95% Confidence Interval); unit: Months, estimated using the Kaplan-Meier
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Months, estimated using the Kaplan-Meier | 30.4 [17.7 to NA] — The upper limit for the 95% CI for median OS and PFS was not reached

5. Secondary Outcome: Overall Survival (OS)
Description: OS will be estimated using the Kaplan-Meier method.
Time Frame: Up to 44 months post radiation
Measure: Median (95% Confidence Interval); unit: Months, estimated using the Kaplan-Meier
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Months, estimated using the Kaplan-Meier | 37.9 [25.4 to NA] — The upper limit for the 95% CI for median OS and PFS was not reached

6. Secondary Outcome: Fatigue as Measured by The Multidimensional Fatigue Inventory (MFI)
Description: Fatigue will be assessed before and after radiotherapy. The Multidimensional Fatigue Inventory (MFI) is a comprehensive self-report instrument designed to measure fatigue. It consists of 20 items rated on a 7-point scale and covers dimensions such as General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Motivation, and Reduced Activity. Each question is score on a 1 to 5 scale, with 1 being 'yes, that is true' and 5 being 'No, that is not true'. The minimum score is 20 and the maximum score is100. The higher the score indicates fatigue.
Time Frame: Pre-radiation on day 1, Last Day of radiation (5-10 days), 1 month post radiation, and 3 months post radiation, change last day of radiation, change 1 month post radiation, change 3 months post radiation
Population: Not all patients completed the measure at every timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Scores on a scale
  Pre-radiation | 55 (16.4)
  Last Day of radiation: number analyzed (Participants) | 34
  Last Day of radiation | 53.6 (13.8)
  1-month post radiation: number analyzed (Participants) | 35
  1-month post radiation | 54.0 (16.6)
  3-month post radiation: number analyzed (Participants) | 33
  3-month post radiation | 52.3 (15.9)
  Change (Last Day of Radiation - Pre-radiation): number analyzed (Participants) | 34
  Change (Last Day of Radiation - Pre-radiation) | 0.1 (11.5)
  Change (1-month post radiation - Pre-radiation): number analyzed (Participants) | 35
  Change (1-month post radiation - Pre-radiation) | -0.4 (15.2)
  Change (3-month post radiation - Pre-radiation): number analyzed (Participants) | 33
  Change (3-month post radiation - Pre-radiation) | -1.4 (12.7)

7. Secondary Outcome: Quality of Life as Measured by Short Form Health Survey (SF-36)
Description: Quality of life will be assessed before and after radiotherapy. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) Each scale is the weighted sum of the questions in their section and are directly transformed into a 0-100 scale i.e., the minimum score is 0, maximum is 100 A higher score indicates less disability Total score on the SF-36 is the summation of all the eight scales
Time Frame: as for outcome 6
Population: Not all patients completed the measure at every timepoint.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Radiation, Palbociclib, Hormone Therapy
Number analyzed (Participants) | 36
Scores on a scale
  Pre-radiation | 41.8 (8.8)
  Last Day of radiation | 42.0 (8.2)
  1-month post radiation | 44.0 (8.1)
  3-month post radiation: number analyzed (Participants) | 35
  3-month post radiation | 44.0 (8.2)
  Change (Last Day of radiation - Pre-radiation) | 0.2 (4.7)
  Change (1-month post radiation - Pre-radiation) | 2.1 (6.6)
  Change (3-month post radiation - Pre-radiation): number analyzed (Participants) | 35
  Change (3-month post radiation - Pre-radiation) | 1.9 (7.3)

8. Secondary Outcome: Quality of Life as Measured by European Organization for Research and Treatment of Cancer Metastases Module (EORTC QLQ-BM22)
Description: Quality of life will be assessed before and after radiotherapy.
  EORTC QLQ-BM22 measures four multi-item scales: painful sites, functional interference, painful characteristics, and psychosocial aspects Each item is scaled from 1 (not at all) to 4 (very much) and directly transformed into a 0-100 scale A higher score in symptom scales indicates greater distress. A higher score in functional scales indicates greater functional ability
Time Frame: as for outcome 6
Population: Not all patients completed the measure at every timepoint.
Measure: Mean (Standard Deviation); unit: EORT QLQ-BM22 score
Groups:
- Treated, Painful Site: Evaluable, Painful Site
- Treated, Pain Characteristics: Evaluable ,Pain Characteristics
- Treated, Functional Interference: Evaluable, Functional Interference
- Treated, Psychological Aspects: Evaluable, Psychological Aspects
Arm/Group | Treated, Painful Site | Treated, Pain Characteristics | Treated, Functional Interference | Treated, Psychological Aspects
Number analyzed (Participants) | 36 | 36 | 36 | 36
EORT QLQ-BM22 score
  Pre-radiation | 28.0 (21.0) | 31.2 (26.5) | 63.6 (30.9) | 61.0 (20.9)
  Last Day of radiation | 21.5 (20.0) | 25.0 (23.7) | 73.4 (25.8) | 68.4 (19.8)
  1-month post radiation | 18.5 (15.1) | 22.2 (24.6) | 74.1 (26.6) | 69.9 (21.7)
  3-month post radiation: number analyzed (Participants) | 35 | 35 | 35 | 35
  3-month post radiation | 17.7 (14.4) | 18.1 (16.6) | 74.8 (21.0) | 68.1 (23.3)
  Change (Last Day of radiation - Pre-radiation) | -6.5 (14.1) | -6.2 (19.4) | 9.8 (18.7) | 7.4 (18.7)
  Change (1-month post radiation - Pre-radiation) | -9.4 (15.7) | -9.0 (25.9) | 10.5 (29.8) | 9.0 (17.1)
  Change (3-month post radiation - Pre-radiation): number analyzed (Participants) | 35 | 35 | 35 | 35
  Change (3-month post radiation - Pre-radiation) | -10.7 (15.8) | -13.7 (20.0) | 11.9 (23.1) | 6.7 (19.0)

9. Secondary Outcome: Quality of Life as Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 15 for Palliative Care (EORTC QLQ-C15-PAL)
Description: Quality of life will be assessed before and after radiotherapy. The EORTC QLQ-C15-PAL measures seven scales: physical functioning, global health status, emotional functioning, fatigue, nausea/vomiting, appetite loss, and constipation For questions 1-14, each item is scaled from 1 (not at all) to 4 (very much) . For question 15 (global QoL), patients respond to a seven-point numerical scale from 1 (very poor overall) to 7 (excellent overall). The scale is scored from 0 to 100. A higher score in symptom scales indicates greater distress.
  A higher score in functional scales indicates greater functional ability. A higher score in global health status indicates a high quality of life.
  Each subscore is computed using the Addendum to the EORTC QLQ-C30 Scoring Manual: Scoring of the EORTC QLQ-C15-PAL.
Time Frame: as for outcome 6
Population: Not all patients completed the measure at every timepoint.
Measure: Mean (Standard Deviation); unit: EORTC QLQ-C15-PAL score
Groups:
- Evaluable, Global Health: Evaluable, Global Health
- Evaluable, Pain: Evaluable Pain
Arm/Group | Evaluable, Global Health | Evaluable, Pain
Number analyzed (Participants) | 36 | 36
EORTC QLQ-C15-PAL score
  Pre-radiation | 72.7 (19.6) | 42.6 (28.9)
  Last Day of radiation | 68.1 (20.5) | 32.4 (28.4)
  1-month post radiation | 72.7 (20.4) | 28.7 (23.8)
  3-month post radiation: number analyzed (Participants) | 35 | 35
  3-month post radiation | 71.9 (20.5) | 28.6 (23.8)
  Change (Last Day of radiation - Pre-radiation) | -4.6 (21.3) | -10.2 (25.3)
  Change (1-month post radiation - Pre-radiation) | 0.0 (22.9) | -13.9 (27.7)
  Change (3-month post radiation - Pre-radiation): number analyzed (Participants) | 35 | 35
  Change (3-month post radiation - Pre-radiation) | -0.5 (19.6) | -13.8 (26.0)

10. Secondary Outcome: Depression as Measured by Hospital Anxiety and Depression Scale (HADS)
Description: Depression will be assessed before and after radiotherapy. The Hospital Anxiety and Depression Scale (HADS) is a 14-item tool used to screen for anxiety and depression, which commonly coexist. The HADS produces a subscale for anxiety (HADS-A) and a separate subscale for depression (HADS-D). The respondent rates each item on a 4-point scale ranging from 0 (absence) to 3 (extreme presence). The total score is out of 42, (21 per subscale) and the range is 0-42. Scores are derived by summing responses for each of the two subscales or for the scale as a whole. Higher scores indicate greater levels of anxiety or depression. The total HADS score may be regarded as a global measure of psychological distress.
Time Frame: as for outcome 6
Population: Not all patients completed the measure at every timepoint.
Measure: Mean (Standard Deviation); unit: HADS score, both depression and anxiety
Groups:
- Evaluable Depression: Evaluable, Depression
- Evaluable Anxiety: Evaluable, Anxiety
Arm/Group | Evaluable Depression | Evaluable Anxiety
Number analyzed (Participants) | 36 | 36
HADS score, both depression and anxiety
  Pre-radiation | 4.9 (3.5) | 6.1 (3.6)
  Last day of radiation | 4.6 (3.5) | 5.3 (3.8)
  1-month post radiation | 4.3 (3.5) | 5.2 (3.6)
  3-month post radiation: number analyzed (Participants) | 34 | 34
  3-month post radiation | 4.1 (3.5) | 5.3 (4.0)
  Change (Last day of radiation - Pre-radiation) | -0.3 (2.0) | -0.8 (1.9)
  Change (1-month post radiation - Pre-radiation) | -0.6 (2.6) | -0.8 (2.3)
  Change (3-month post radiation - Pre-radiation): number analyzed (Participants) | 34 | 34
  Change (3-month post radiation - Pre-radiation) | -0.7 (3.5) | -0.8 (3.0)

11. Secondary Outcome: Number of Participants With Adherence as Measured by Drug Diary
Description: Adherence will be determined by number of days drug taken divided by number of days drug should have been taken over the time period of the study.
Time Frame: as for outcome 6
Population: At each timepoint, there are a different number of patients analyzed due to missing data, patients that were lost to follow up or removed due to disease progression.
Measure: Count of Participants; unit: Participants
Groups:
- Evaluable Palbo: Evaluable, Palbo
- Evaluable Hormone: Evaluable, Hormone therapy
Arm/Group | Evaluable Palbo | Evaluable Hormone
Number analyzed (Participants) | 36 | 36
Participants
  Pre-radiation | 36 | 36
  Last Day of radiation: number analyzed (Participants) | 36 | 35
  Last Day of radiation | 33 | 35
  1-month post radiation: number analyzed (Participants) | 34 | 33
  1-month post radiation | 25 | 29
  3-month post radiation: number analyzed (Participants) | 31 | 30
  3-month post radiation | 26 | 30

ADVERSE EVENTS:
Time Frame: All-Cause Mortality monitored/assessed up to 44 months. Adverse Events were monitored/assessed up to 3 months post Radiation Therapy.
Groups:
- Grade 1 Adverse Event; Grade 2 Adverse Event; Grade 3 Adverse Event; Grade 4 Adverse Event; Grade 5 Adverse Event: Patients undergo radiation therapy over 5-10 days and receive palbociclib PO QD on days 1-21. At the discretion of treating physician, patients also receive letrozole, anastrozole, exemestane, or tamoxifen PO QD on days 1-28, or fulvestrant IM on days 1 and 15 of cycle 1 and on day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Anastrozole: Given PO
  Exemestane: Given PO
  Fulvestrant: Given IM
Arm/Group | Grade 1 Adverse Event | Grade 2 Adverse Event | Grade 3 Adverse Event | Grade 4 Adverse Event | Grade 5 Adverse Event
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 7/36
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/36 | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 31/36 | 30/36 | 17/36 | 2/36 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grade 1 Adverse Event (N=36) | Grade 2 Adverse Event (N=36) | Grade 3 Adverse Event (N=36) | Grade 4 Adverse Event (N=36) | Grade 5 Adverse Event (N=36)
Anemia (Blood and lymphatic system disorders) | 12 | 2 | 0 | 0 | 0
Anorexia (General disorders) | 2 | 0 | 0 | 0 | 0
Bilateral Arm Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Bilateral Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 0
Dry Skin/Rash on Back (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Dyspnea (General disorders) | 1 | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 11 | 5 | 0 | 0 | 0
Gastroesophagealreflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lymphocyte Count Decrease (Blood and lymphatic system disorders) | 2 | 8 | 7 | 2 | 0
Mouth Sores (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neutrophil Count Decrease (Blood and lymphatic system disorders) | 7 | 9 | 13 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Platelet Count Decreased (Investigations) | 8 | 2 | 0 | 0 | 0
Pruitus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Skin Desquamation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 0 | 0
Weight Loss (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
White Blood Cell Decrease (Investigations) | 9 | 17 | 12 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Moderate erythema over sternum (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Any Grade 4 AE - excluding neutropenia and leukpenia (Investigations) | 0 | 0 | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT03691493/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT03691493/ICF_000.pdf